CLINICAL TRIAL: NCT04631263
Title: A Randomized, Evaluator-blinded, Parallel Group, no Treatment Controlled, Multi-center Study to Evaluate Effectiveness and Safety of GP0109 for Augmentation and Correction of Retrusion in the Chin Region
Brief Title: New Dermal Filler for Chin Correction and Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43BBJ2001
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-06

CONDITIONS: Chin Augmentation and Correction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Device: Hyaluronic Acid
- Control Group (No Intervention)

INTERVENTIONS:
Device: Hyaluronic Acid — Injectable gel. Chin correction and augmentation for retrusion
  Other Names: GP0109
  Arms: Treatment Group

SUMMARY:
Randomized, evaluator-blinded, no treatment controlled multicenter study to evaluate safety and effectiveness of GP0109 for augmentation and correction or retrusion in the chin region in Canada

ELIGIBILITY:
Inclusion Criteria:

* subject willing to comply with the requirements of the study
* subject intent to receive treatment for augmentation and correction of retrusion in the chin region
* subject with mild or moderate (grade 1 or 2) on the GCRS

Exclusion Criteria:

* subjects presenting with know allergy to HA (hyaluronic acid) filler or amide local anesthetics
* subjects with any previous facial surgery below the nasal line or previous HA filler or collagen below the nasal line within 12 months
* subjects in any other interventional clinical study within 30 days before baseline

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Responder rate based on the Galderma Chin Retrusion Scale as assessed live by the Blinded Evaluator | 3 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (6):
- Canada (6):
  - Galderma Research Site, Calgary, Alberta
  - Galderma Research Site, Vancouver, British Columbia
  - Galderma Research Site, Burlington, Ontario
  - Galderma Research Site, Toronto, Ontario
  - Galderma Research Site, Woodbridge, Ontario
  - Galderma Research Site, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: No